CLINICAL TRIAL: NCT07393412
Title: PRIME (Precision Registry for Integrated Cardio-cerebrovascular Medicine & Evidence)
Brief Title: Identifying Risk Factors and Predicting Future Health Outcomes for Korean Patients With Heart and Blood Vessel Diseases: A Long-term Follow-up Study
Status: Not yet recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: SMC IRB 2025-12-061
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Diseases (CVD); Cerebro Vascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Years

INTERVENTIONS:
Drug: Standard Medical Therapy — Routine pharmacological treatments including antiplatelets, antihypertensives
Procedure: Revascularization Procedures — Surgical or interventional procedures such as PCI (Percutaneous Coronary Intervention) or stent thrombectomy for stroke.
Behavioral: Lifestyle Modification — Habitual factors including smoking cessation, physical activity, and dietary habits monitored during the follow-up.

SUMMARY:
This study aims to establish a comprehensive, long-term clinical registry infrastructure for heart and brain vascular diseases (cardiovascular diseases and stroke) at Samsung Medical Center. In South Korea, these diseases are a leading cause of death, with a rapidly increasing burden due to an aging population and changing lifestyles. Despite this, there is a lack of large-scale, systematic data specifically focused on the long-term clinical course and unique characteristics of Korean patients.

The central hypothesis of this study is that the establishment of a standardized registry infrastructure-integrating both retrospective (historical) and prospective (future) data collection-will provide a more accurate and comprehensive understanding of the natural history and risk factors of heart and brain vascular diseases in the Korean population than currently available fragmented data. By combining existing medical records with ongoing patient follow-up, this infrastructure will serve as a critical scientific platform for developing personalized prevention and precision medicine strategies.

By building this organized data collection system, the study will:

Construct a robust infrastructure to collect uniform, high-quality clinical data, encompassing both past medical history (retrospective) and future clinical progress (prospective) from a large population of Korean patients.

Monitor long-term health outcomes and the progression of diseases by tracking patients over many years.

Analyze the interaction between various risk factors and patient outcomes to identify population-specific patterns.

Create a scalable platform that can integrate advanced technologies, such as multi-omics and digital health tools, for future research.

Ultimately, this integrated registry infrastructure is expected to provide the essential scientific evidence needed to optimize clinical guidelines and improve the long-term quality of life for patients with heart and brain vascular diseases in Korea.

ELIGIBILITY:
Inclusion Criteria:

A patient who visited Samsung Medical Center due to cardiovascular and cerebrovascular disease.

Exclusion Criteria:

A patient deemed unable to participate in the study based on the judgment of the medical staff.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients diagnosed with or treated for heart and brain vascular diseases (cardiovascular diseases and stroke) at Samsung Medical Center, a tertiary academic hospital in Seoul, Korea.
  This cohort includes:
  Retrospective Group: Patients with clinical records within the hospital's historical database to analyze past clinical courses and long-term outcomes.
  Prospective Group: Patients newly visiting or currently under follow-up care at the heart, stroke, and vascular centers who consent to long-term monitoring.
  The population covers a wide clinical spectrum, from acute emergency cases (e.g., myocardial infarction, ischemic stroke) to chronic management.
Sampling Method: Probability Sample
Enrollment: 800000 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-11-27 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Major Adverse Cardio-Cerebrovascular Events (MACCE) | Up to 20 years (from the date of enrollment until the end of the follow-up period)